CLINICAL TRIAL: NCT00682617
Title: Hip Osteoarthritis: Effects of Structured Exercise Programs on Pain and Long-term Disability
Brief Title: Hip Osteoarthritis: Effects of Exercise Programs on Pain and Disability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Nels Carlson, MD, Oregon Health and Science University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: IRB #290
Record Dates: First submitted 2008-05-20; First posted 2008-05-22 (Estimated); Results first posted 2020-03-24 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Hip Osteoarthritis
Keywords: hip; osteoarthritis; exercise; disability; physical function
MeSH Terms: conditions — Osteoarthritis, Hip; Osteoarthritis; Motor Activity | interventions — Waiting Lists

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Waitlist Control (Experimental): Delayed intervention. 3 months on waitlist, crossover to intervention (3 additional months)
  Interventions: Behavioral: Waitlist, delayed intervention
- 3 Month Exercise Program (Experimental): 3 month exercise program
  Interventions: Behavioral: Structured exercise program

INTERVENTIONS:
Behavioral: Structured exercise program — Exercise intervention will consist of a three-month, supervised, facility-based, hip-specific strengthening, flexibility, and endurance exercise program. The intervention will consist of two phases and take place at OHSU rehabilitation services. Phase 1 will be a two-week orientation and general conditioning program. Phase 2 will be a ten-week progressive workload program. Subjects in both Phase 1 and Phase 2 will meet two to three times per week for 45 minutes per session. Phase 1 will be group sessions with more individualized orientation and attention by the exercise instructors. Phase 2 will begin progressive conditioning and utilize exercise groups of four to six subjects.
  Other Names: Group 2
  Arms: 3 Month Exercise Program
Behavioral: Waitlist, delayed intervention — Due to limited space in exercise intervention classes, subjects may be placed on a waitlist for 3 months. When an opening becomes available, the subject will begin the exercise program identical to that of Group 2
  Other Names: Group 1
  Arms: Waitlist Control

SUMMARY:
Osteoarthritis is the most common form of arthritis in the United States. It is estimated that 20 million Americans have arthritis, and the annual societal cost is $95 billion. Several exercise studies have shown modest improvements in disability, physical performance, and pain in subjects with knee osteoarthritis. While similar results have been suggested in hip osteoarthritis, well-designed randomized clinical trials have not been conducted. Exercise programs appear beneficial but without adherence, the beneficial effects of exercise for knee and hip osteoarthritis decline over time. A well-designed, evidence-based, arthritis-specific study controlling for exercise duration, frequency and adherence is needed. The objective of this study is to determine the effects of structured exercise programs on self-reported pain and disability in adults with hip osteoarthritis. This prospective, randomized study with a wait-list control is designed to develop preliminary data to support an R01 funding request for a large, randomized clinical trial. All exercise interventions and outcome assessments will take place at OHSU in the Orthopaedics and Rehabilitation Clinics, Rehabilitation Services physical therapy gym, and the General Clinical Research Center. Subjects will be selected to include individuals representative of the larger population with documented hip osteoarthritis. This three-month study will evaluate the effects of an aerobic and resistance exercise program on pain and disability in individuals with hip osteoarthritis. Outcome assessment will follow the Outcome Measures in Rheumatology (OMERACT) recommendations for a core set of outcome measures for clinical trials in arthritis and assess pain, physical function, patient global assessment, and joint imaging. Data analysis will focus on comparing pre- and post-intervention endpoints using conventional statistical analyses such as repeated-measure analysis of variance for repeated continuous measures (e.g. walking distance), and non-parametric methods such as Chi-square or frequency analysis for proportions (e.g. visual pain scores).

ELIGIBILITY:
Inclusion Criteria:

* Age 21 years or more
* Pain at least once a week in one or both hips
* Difficulty with at least one of the following secondary to hip pain: walking 1/4 mile, climbing stairs, getting in and out of a car, rising from a chair, lifting and carrying groceries, getting out or bed, getting out of the bathtub, or performing shopping, cleaning or self-care activities
* Radiographic evidence of femoral and/or acetabular osteophytes on radiograph -OR- radiographic evidence of axial joint space narrowing and active hip flexion </= 115 degrees
* Primary care physician's written consent to participate in the exercise-based protocol. If te subject does not have a primary care physician, the subject will complete a screening questionnaire for coronary artery disease. If the subject screens as "high risk", te subject will be excluded from the study

Exclusion Criteria:

* A medical condition that precludes safe participation in an exercise program including active cardiac disease, angina, class III heart failure, myocardial infarction in the past year
* Screening as "high risk" for coronary artery disease
* Inflammatory arthritis (e.g. psoriatic or rheumatoid)
* Collecting workers' compensation
* Involved in litigation regarding pain and/or disability
* Unable to walk six minutes without cane or assistive device
* Participating in a conflicting research study
* Significant, symptomatic knee or ankle osteoarthritis
* Other lower extremity pathology including peripheral vascular disease that would preclude participation in an exercise program
* Pregnancy

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2007-05-23 (Actual); Primary Completion 2010-11-11 (Actual); Study Completion 2010-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nels Carlson, M.D., Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University Center for Health & Healing, Portland, Oregon, United States

REFERENCES:
- [Background] Thompson AR, Christopherson Z, Marshall LM, Carlson HL, Carlson NL. A Pilot Randomized Controlled Trial for Aerobic and Strengthening Exercises on Physical Function and Pain for Hip Osteoarthritis. PM R. 2020 Mar;12(3):229-237. doi: 10.1002/pmrj.12262. Epub 2019 Dec 12. PMID 31600429

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Waitlist Control | 3 Month Exercise Program
Started | 13 | 28
Completed | 10 | 21
Not Completed | 3 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Waitlist Control | 3 Month Exercise Program | Total
Number analyzed (Participants) | 10 | 21 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.8 (9.1) | 59.7 (8.7) | 60.1 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 16
  Male | 3 | 12 | 15
6 Minute Walk Test [Median (Inter-Quartile Range); unit: meters] | 538 [493 to 584] | 567 [527 to 678] | 562 [512 to 646]
WOMAC Physical Function Subscale [Median (Inter-Quartile Range); unit: units on a scale] — The WOMAC Physical Function Subscale has a range of 0-68, with higher scores indicating worse functional limitations.
  units on a scale | 21 [17 to 26] | 22 [16 to 25] | 21 [16 to 25]
Pain Visual Analog Scale [Median (Inter-Quartile Range); unit: units on a scale] — Evaluated using a 100mm pain VAS (range 0-100), with higher scores indicating worse pain.
  units on a scale | 37 [33 to 51] | 37 [23 to 46] | 37 [23 to 47]

OUTCOME MEASURES:

1. Primary Outcome: Change in 6-minute Walk Test
Description: Calculated as change from baseline to 3 months
Time Frame: 3 months
Measure: Median (Inter-Quartile Range); unit: meters
Arm/Group | Waitlist Control | 3 Month Exercise Program
Number analyzed (Participants) | 10 | 21
meters | 22 [-10 to 64] | 49 [24 to 83]

2. Secondary Outcome: Change in Pain Visual Analog Scale
Description: Evaluated using a 100mm pain VAS (range 0-100), with higher scores indicating worse pain. Calculated as change from baseline to 3 months.
Time Frame: 3 months
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Waitlist Control | 3 Month Exercise Program
Number analyzed (Participants) | 10 | 21
units on a scale | -3 [-14 to 1] | -5 [-19 to -1]

3. Secondary Outcome: Change in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Physical Function Subscale
Description: The WOMAC Physical Function Subscale has a range of 0-68, with higher scores indicating worse functional limitations. Calculated as change from baseline to 3 months.
Time Frame: 3 months
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Waitlist Control | 3 Month Exercise Program
Number analyzed (Participants) | 10 | 21
units on a scale | -2 [-4 to 2] | -5 [-9 to -2]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over the duration of the intervention (3 months).
Arm/Group | Waitlist Control | 3 Month Exercise Program
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/21
Other Adverse Events (participants affected / at risk) | 0/10 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes